CLINICAL TRIAL: NCT07235306
Title: Ensartinib for the Treatment of Patients With ALK-Mutated Stage III Unresectable NSCLC: A Multicenter, Randomized Controlled, Double-blind Clinical Study
Brief Title: Ensartinib After Chemoradiotherapy in Stage III ALK-Mutated NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yaping Xu, chiefphysician, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L25-616
Record Dates: First submitted 2025-09-23; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage III; Ensartinib; Chemoradiotherapy; ALK
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ensartinib (Experimental): Ensartinib (225mg orally, once daily), in accordance with the randomization schedule
  Interventions: Drug: Ensartinib 225mg
- Placebo Ensartinib (Placebo Comparator): Matching placebo for Ensartinib (225mg orally, once daily), in accordance with the randomization schedule
  Interventions: Drug: Placebo Ensartinib 225mg

INTERVENTIONS:
Drug: Ensartinib 225mg — 225mg once daily, until disease progression, unacceptable toxicity or other discontinuation criteria are met
  Arms: Ensartinib
Drug: Placebo Ensartinib 225mg — 225mg once daily, until disease progression, unacceptable toxicity or other discontinuation criteria are met
  Arms: Placebo Ensartinib

SUMMARY:
The PACIFIC study established the standard of care for immunotherapy consolidation after chemoradiotherapy (CRT) in patients with unresectable stage III non-small cell lung cancer (NSCLC). However, its benefit is limited in patients with driver gene mutations. The LAURA study established a new paradigm of targeted consolidation therapy after CRT for patients with EGFR mutations. Although retrospective data support the efficacy of ALK-TKIs, no randomized controlled trial (RCT) has clearly demonstrated the value of ALK-TKI maintenance therapy after CRT. This study adopts a multicenter, randomized, double-blind, placebo-controlled design aimed at evaluating the efficacy and safety of ensartinib in patients with ALK-positive unresectable stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged at least 18 years
* Histologically or cytologically confirmed Stage III unresectable non-small cell lung cancer (NSCLC) with curative treatment intent
* ALK mutations assessed by FISH, IHC, or NGS
* ECOG Performance Status of 0 or 1
* Completion of platinum-based concurrent or sequential chemoradiotherapy as per protocol requirements
* Chemoradiotherapy must have been completed ≤ 6 weeks prior to randomization
* No disease progression during or after chemoradiotherapy
* Life expectancy > 12 weeks
* Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to initiation of treatment
* Signed informed consent form obtained from the patient or their legally authorized representative
* Male and female patients of childbearing potential agree to use highly effective contraception methods from before entering the trial, throughout the study, and until 8 weeks after discontinuation of study treatment

Exclusion Criteria:

* Mixed histology of small cell and non-small cell lung cancer
* Symptomatic pneumonitis following chemoradiotherapy that has not resolved to ≤ Grade 1 (per CTCAE criteria) prior to randomization;
* Any unresolved toxicity from prior chemoradiotherapy with toxicity ≥ Grade 2 (according to CTCAE criteria);
* Poor cardiac function, including but not limited to any of the following:

  * Mean resting corrected QT interval (QTc) > 470 msec (obtained from 3 ECGs);
  * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG;
  * Any factors that increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or concomitant use of any known drugs that prolong the QT interval and may lead to Torsades de Pointes;
* Inadequate bone marrow reserve or organ function;
* History of other malignant malignancies, except for adequately treated non-melanoma skin cancer or malignant lentigo, cured carcinoma in situ, or other solid tumors cured > 5 years ago with no evidence of disease and considered by the treating physician to have a low risk of recurrence;
* Severe or uncontrolled systemic diseases: including uncontrolled hypertension and active bleeding tendency; or active infections, including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV);
* Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of ensartinib;
* Any prior chemotherapy, radiotherapy, immunotherapy, or investigational drug therapy beyond the definitive treatment for locally advanced disease;
* Prior treatment with any ALK tyrosine kinase inhibitor (ALK-TKI);
* Major surgery within 4 weeks prior to the first dose of study drug;
* Current use of medications known to be strong inducers of CYP3A4 (which cannot be discontinued at least 3 weeks prior to the first dose of study drug);
* Known hypersensitivity to ensartinib or any excipient in this product;
* Pregnant or lactating women;
* History of definite neurological or psychiatric disorders, including epilepsy or dementia;
* Any other condition that, in the judgment of the investigator, would make the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
progressive free survival | From enrollment to the end of treatment, up to 100 months
  disease progression according to RSCIST v1.1 or intolerable toxicity according to CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate | From first dose of study drug until disease progression, assessed up to approximately 12 months
  ORR is defined as the proportion of participants whose best overall response is complete response (CR) or partial response (PR) as assessed by the investigator according to RECIST 1.1
Disease Control Rate | From first dose of study drug until disease progression, assessed up to approximately 12 months
  DCR is defined as the proportion of participants achieving a best overall response of complete response (CR), partial response (PR), or stable disease (SD) as assessed by the investigator according to RECIST 1.1
Overall Survival (OS) | From randomization until death from any cause, up to 120 months
  OS is defined as the time from randomization until death due to any cause.
Central Nervous System Progression-Free Survival (CNS-PFS) | From randomization until CNS progression or death, up to 100 months
  CNS-PFS is defined as the time from randomization to the first documented intracranial progression (as assessed by MRI ) or death from any cause, whichever occurs first.
Incidence of Adverse Events (AEs) | Approximately up to 100 months
  AEs graded by CTCAE version 5.0

OTHER OUTCOMES:
Exploratory Analysis of Biomarkers and Efficacy | Blood samples will be collected at the following time points: before chemoradiotherapy, within 6 weeks after chemoradiotherapy, at 6 months of medication, and through study completion, an average of 5 year
  To explore the correlation between potential biomarkers and efficacy outcomes (PFS/ORR/DCR/OS/CNS-PFS) through analysis of blood samples